CLINICAL TRIAL: NCT07300046
Title: A Randomized Study to Assess the Tolerability Profile of Two Concentrations of Liquid Metformin (100 mg/mL and 250 mg/mL) Compared With Standard Metformin Tablets
Brief Title: Tolerability Study of Liquid Metformin (100 and 250 mg/mL) vs IR Tablets
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Aspargo Labs, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: ASP-019-Met
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-Arm Crossover (Experimental)
  Interventions: Drug: Liquid Metformin 100 mg/mL; Drug: Liquid Metformin 250 mg/mL; Drug: Standard Metformin Immediate-Release Tablet

INTERVENTIONS:
Drug: Liquid Metformin 100 mg/mL — A single oral dose of a liquid metformin formulation at a concentration of 100 mg/mL will be administered under fasting conditions in one period of the crossover to assess tolerability and safety.
Drug: Liquid Metformin 250 mg/mL — A single oral dose of a liquid metformin formulation at a concentration of 250 mg/mL will be administered under fasting conditions in one period of the crossover to assess tolerability and safety.
Drug: Standard Metformin Immediate-Release Tablet — A single oral dose of standard immediate-release metformin tablet(s) will be administered under fasting conditions in one period of the crossover to assess tolerability and safety.

SUMMARY:
This is an open-label, randomized study evaluating the tolerability of two concentrations of liquid metformin formulations (100 mg/mL and 250 mg/mL) compared with standard immediate-release metformin tablets in healthy adult subjects. Each participant will receive single oral doses of study treatments in a randomized sequence. Safety and tolerability will be assessed through adverse event monitoring, gastrointestinal symptom evaluations, vital signs, clinical laboratory tests, and ECGs.

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults 18 to 55 years of age, inclusive.

Body mass index (BMI) between 18.0 and 30.0 kg/m², inclusive.

Medically healthy based on medical history, physical examination, vital signs, clinical laboratory evaluations, and 12-lead ECG, in the opinion of the investigator.

Non-smoker or light smoker (10 cigarettes per day or fewer, or equivalent) willing to abstain during study confinement periods.

Able to provide written informed consent before any study-specific procedures are conducted.

Willing and able to comply with all study requirements, including fasting, dosing restrictions, and safety/tolerability assessments.

Females of childbearing potential must use acceptable contraception as determined by the investigator.

Exclusion Criteria:

* Known hypersensitivity or contraindication to metformin or any excipients in the study formulations.

History or presence of clinically significant cardiovascular, hepatic, renal, gastrointestinal, endocrine, hematologic, neurologic, or psychiatric disease that, in the investigator's opinion, could interfere with participation or data interpretation.

Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73 m², or any clinically significant abnormal clinical laboratory findings.

Prior history of lactic acidosis.

Current or recent (within 14 days before first dose) use of prescription drugs, over-the-counter medications, herbal products, or dietary supplements, unless approved by the investigator.

Positive test for hepatitis B surface antigen, hepatitis C antibody, or HIV.

Positive urine drug screen or positive alcohol breath test at screening or at check-in.

Participation in another clinical trial or receipt of an investigational drug or device within 30 days or 5 half-lives (whichever is longer) before first study dose.

Donation of ≥450 mL of blood, or significant blood loss, within 8 weeks before the first study dose.

Pregnant or breastfeeding females.

Women of childbearing potential not using acceptable contraception.

Any condition or finding that, in the opinion of the investigator, would make the subject unsuitable for the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-06-15 (Estimated); Primary Completion 2026-08-15 (Estimated); Study Completion 2026-08-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Gastrointestinal Treatment-Emergent Adverse Events (GI TEAEs) | From each study dose through 24 hours postdose in each treatment period
Severity of Gastrointestinal Treatment-Emergent Adverse Events | From each study dose through 24 hours postdose in each treatment period

IPD SHARING:
Plan to Share IPD: No